CLINICAL TRIAL: NCT01942876
Title: Preventing Drug Use in Low Income Clinic Populations
Acronym: QUIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DESPR DA022445
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Drug Use; Harmful Use
Keywords: Drugs; at risk; community health center patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The Quit Using Drugs Intervention Trial (QUIT) experimental arm includes: screening, very brief clinician advice, and telephone drug-use health education to reduce 'at risk' drug use and thus interrupt progression from casual or episodic abuse to dependence.
  Interventions: Behavioral: Quit Using Drugs Intervention Trial
- Control (Sham Comparator): This arm will receive a sham telephone intervention of equivalent duration on health behavior maintenance.
  Interventions: Behavioral: Health behavior maintenance

INTERVENTIONS:
Behavioral: Quit Using Drugs Intervention Trial — The goal of the Quit Using Drugs Intervention Trial (QUIT) is to conduct a small RCT of a primary care clinic-based very brief intervention protocol for reducing the use of illegal drugs and the occurrences of drug-related harm in low-income, racially-diverse patient populations at two 'safety-net' clinics in Los Angeles. The design will emphasize screening, very brief clinician advice, and telephone drug-use health education to reduce 'at risk' drug use and thus interrupt progression from casual or episodic abuse to dependence.
  Other Names: QUIT
  Arms: Intervention
Behavioral: Health behavior maintenance — This attention-control arm will receive a sham telephone intervention of equivalent duration on health behavior maintenance.
  Other Names: Attention-Control condition
  Arms: Control

SUMMARY:
The proposed study will address the critical need to reduce illegal drug use, in particular drug use, and the occurrence of drug-related harm in low-income racially diverse patient populations at urban primary care safety-net clinics. Since they are at risk for accelerated trajectories to drug dependence once drug use begins, low-income racially diverse populations pose particular concern for public health policy makers and drug-use prevention efforts. The study will be the first to standardize drug screening and primary-care clinician delivered brief intervention among racially diverse "at risk" drug users, that is users with casual or frequent use without the physiological or psychological manifestations of dependence, to reduce their 'at risk' use of drugs, and it may effectively interrupt their pathway to dependence.

DETAILED DESCRIPTION:
The Quit Using Drugs Intervention Trial (QUIT) will be the first randomized controlled trial in the U.S. that is powered to detect the effect of a primary care clinician delivered brief intervention protocol for reducing 'at risk' drug use and drug-related harm among low-income adult patients (ages 18 and older) at multiple safety net clinics in Los Angeles County. For this small trial, we will sample patients with 'at risk' use of drugs (marijuana, crack/cocaine, amphetamines/methamphetamines, inhalants, sedatives or sleeping pills, hallucinogens, and opiates), the most commonly used serious drugs among patients at our clinic sites. "At risk" drug use is defined in this study as current use (past 90 days) of drug measured as a self-reported total score of 4 to 26 on the WHO Alcohol Substance Involvement Screening Test (ASSIST). A total of 7,000-8,000 patients will be approached for screening to yield a 3-month effective sample size of 245 eligible patients per condition (1) an intervention condition involving drug use health education or (2) a control condition involving care as usual. In the intervention condition, very brief (less than 5 minutes) clinician advice regarding quitting drug use will be followed by two 2 and 6 week post-visit drug health education sessions on quitting drug use and cautioning against use of other 'at risk' substance use such as alcohol and tobacco. Patients assigned to the control condition will receive standard care for drug use at the baseline visit with their clinician. Follow-up assessments will be conducted at 3 month post-randomization. The framework for the QUIT project is the Social Action Theory, and the brief intervention protocol is based on NIDA's principles on prevention research and the utility of the 5 A's approach for assisting behavioral changes among patients (Ask, Advise, Assess, Assist, Arrange) in the clinic setting. If found to be effective in the community health center setting, this clinician and telephone drug-use health education program could become a model for health promotion activities. that would be expanded to all 'at risk' substance use and shared between community health centers.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and older
* report of drug use in the previous 90 days (i.e., (marijuana, crack/cocaine, amphetamines/methamphetamines, inhalants, sedatives or sleeping pills, hallucinogens, and opiates)
* an ASSIST score between 4 and 26 indicating 'at risk' drug use
* English or Spanish speaking
* able (not cognitively impaired) and willing to cooperate with data collection and research procedures, including 2 telephone counseling sessions and 3 month follow-up assessments

Exclusion Criteria:

* Pregnant
* Drug or alcohol dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Self-reported number of drug-free days at 3 month | past 30 and 90 days

SECONDARY OUTCOMES:
Decrease in drug-related harm (e.g., unemployment and job absenteeism, poor social support, poor health-related quality of life, HIV risk behaviors, motor vehicle accidents, and inpatient health services utilization). | 6 and 12 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Gelberg, MD, MSPH, Principal Investigator — UCLA Department of Family Medicine
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Gelberg L, Andersen RM, Afifi AA, Leake BD, Arangua L, Vahidi M, Singleton K, Yacenda-Murphy J, Shoptaw S, Fleming MF, Baumeister SE. Project QUIT (Quit Using Drugs Intervention Trial): a randomized controlled trial of a primary care-based multi-component brief intervention to reduce risky drug use. Addiction. 2015 Nov;110(11):1777-90. doi: 10.1111/add.12993. PMID 26471159
- [Result] Baumeister SE, Gelberg L, Leake BD, Yacenda-Murphy J, Vahidi M, Andersen RM. Effect of a primary care based brief intervention trial among risky drug users on health-related quality of life. Drug Alcohol Depend. 2014 Sep 1;142:254-61. doi: 10.1016/j.drugalcdep.2014.06.034. Epub 2014 Jul 4. PMID 25042213
- [Derived] Bone CW, Goodfellow AM, Vahidi M, Gelberg L. Prevalence of Sexual Violence and its Association with Depression among Male and Female Patients with Risky Drug Use in Urban Federally Qualified Health Centers. J Urban Health. 2018 Feb;95(1):111-115. doi: 10.1007/s11524-017-0213-7. PMID 29340911